CLINICAL TRIAL: NCT06816303
Title: Adult Patients With Diabetes Mellitus, on Drug Treatment, on the List or Already Undergoing Orthotopic Liver Transplantation: an Observational Study
Brief Title: Patients With Diabetes Mellitus on Drug Treatment on the List or Already Undergoing Orthotopic Liver Transplantation
Acronym: DiaBoLT2021
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DiaBoLT2021
Record Dates: First submitted 2024-11-28; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus Type 2; Liver Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
observational study through which we aim to collect information on metabolic compensation, the degree of satisfaction with hypoglycemic therapy, the onset of complications of diabetes or liver disease, evaluation of survival, in patients on the list for at least three months or already undergoing liver transplantation for at least three months

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* presence on the list for OLT for at least 3 months or have already been submitted to OLT for at least 3 months
* age ≥ 18 years
* signature of written informed consent to participate in the observational study, either by the participant or legal guardian

Exclusion Criteria:

- Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients followed for hepatological problems on the list for OLT or post-transplant with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
glycosilated hemoglobin (%) | through study completion, an average of 5 years
  glycometabolic control in relation to therapy

SECONDARY OUTCOMES:
degree of satisfaction with therapy | through study completion, an average of 5 years
  degree of satisfaction with therapy through the administration of Diabetes Treatment Satisfaction Questionnaire (DTSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Brodosi, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Lucia Brodosi, Bologna, BO, Italy